CLINICAL TRIAL: NCT05201794
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Double-dummy, Multicenter Trial Assessing the Efficacy and Safety of Two Dose Regimens of JNJ-64281802 for the Prevention of Dengue Infection
Brief Title: A Study of JNJ-64281802 for the Prevention of Dengue Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to portfolio reprioritization. This decision is not based on any safety concerns.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR109157; 64281802DNG2004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-01-10; First posted 2022-01-21 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High-dose JNJ-64281802 regimen (HDR) (Experimental): Participants will receive JNJ-64281802 400 milligrams (mg) loading dose (LD) twice daily for 48 hours (2 days), followed by JNJ-64281802 150 mg maintenance dose (MD) once daily for 26 days in fed conditions.
  Interventions: Drug: JNJ-64281802
- Low-dose JNJ-64281802 regimen (LDR) (Experimental): Participants will receive JNJ-64281802 150 mg LD twice daily for 48 hours (2 days), followed by JNJ-64281802 50 mg MD once daily for 26 days in fed conditions.
  Interventions: Drug: JNJ-64281802
- Placebo (Placebo Comparator): Participants will receive JNJ-64281802 matching placebo LD and MD from Day 1 to Day 28.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-64281802 — JNJ-64281802 tablets will be administered orally as per the defined regimens.
  Arms: High-dose JNJ-64281802 regimen (HDR); Low-dose JNJ-64281802 regimen (LDR)
Drug: Placebo — Matching placebo for each dose level as tablet will be administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the prophylactic effect of JNJ-64281802 with respect to the prevention of laboratory-confirmed dengue virus (DENV) infection up to the last day of dosing among participants who have no evidence of current DENV infection at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, and vital signs performed at screening. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities to be not clinically relevant. This determination must be recorded in the participant's source documents
* Must have a body mass index (BMI, weight in kilogram [kg] divided by the square of height in meters) between 18.0 and 35.0 kilograms per meter square (kg/m^2) inclusive, and a body weight of greater than or equal to (>=) 40.0 kg at screening
* A woman must have a negative highly sensitive urine pregnancy test at screening
* A male participant must agree not to donate sperm for the purpose of reproduction during the study and for >= 90 days after receiving the last dose of study intervention
* Must sign an informed consent form (ICF) (or their legally acceptable representative must sign) indicating that the participant understands the purpose of, and procedures required for, the study and is willing to participate in the study

Exclusion Criteria:

* Having any dengue virus (DENV)-associated clinical signs and symptoms
* Known allergies, hypersensitivity, or intolerance to JNJ-64281802 or its excipients
* Any clinically relevant skin disease (as assessed by the investigator) in the past 3 months such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, and urticaria
* Reduced immune function to be: (a) Known or suspected congenital or acquired immunodeficiency; or (b) receipt of immunomodulation therapy within the last 6 months (such as anticancer chemotherapy or radiation therapy)
* Received an investigational intervention (including investigational vaccines other than a corona virus disease 2019 [COVID-19] vaccine) or used an invasive investigational medical device within 3 months before the planned first dose of study intervention or received an investigational biologic product within 3 months prior to enrollment or 5 half-lives, whichever is longer, before the planned first dose of study intervention, or is currently enrolled in an investigational study

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1595 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (38):
- Brazil (11):
  - Universidade Federal De Minas Gerais - Hospital das Clínicas, Belo Horizonte
  - HUJM - UFMT - Hospital Universitário Júlio Müller - Universidade Federal do Mato Grosso, Cuiabá
  - Hospital e Maternidade Sao Joao de Deus, Laranjeiras do Sul
  - Fundacao De Medicina Tropical Doutor Heitor Vieira Dourado, Manaus
  - Fundacao Universidade Federal de Mato Grosso do Sul, Mato Grosso Do Sul
  - Policlínica Regional Dr Sérgio Arouca, Niterói
  - UPA Unidade de Pronto Atendimento Mário Monteiro, Niterói
  - Instituto de Pesquisas em Patologias Tropicais de Rondônia - IPEPATRO, Porto Velho
  - Centro Bangu - Centro Municipal de Saude Waldyr Franco, Rio de Janeiro
  - Fundacao Oswaldo Cruz Instituto Nacional de Infectologia Evandro Chagas, Rio de Janeiro
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
- Colombia (8):
  - CAIMED Acacias, Acacías
  - CAIMED Aguazul, Aguazul
  - Centro de Reumatologia y Ortopedia, Barranquilla
  - Hospital Universidad del Norte, Barranquilla
  - Centre of Care and Diagnosis of the Infectious Diseases (CDI), Bucaramanga
  - Centro de Investigaciones Clinicas S A S, Cali
  - Programa de Estudio y Control de Enfermedades Tropicales, Medellín
  - Centro de Atencion e Investigacion Medica S.A. - CAIMED, Yopal - Casanare
- Malaysia (2):
  - Klinik Kesihatan Kuang, Kuang
  - Klinik Kesihatan Pandamaran, Port Klang
- Mexico (4):
  - Centro Medico Jojutla, Jojutla
  - Medical Care & Research SA de CV, Mérida
  - Unidad de Proyectos Clínicos de Oriente UPCO, Valladolid
  - FAICIC S. de R.L. de C.V., Veracruz
- Panama (4):
  - Cevaxin 24 de diciembre, Cuidad de Panama
  - Centro de Vacunacion Internacional CEVAXIN Av Mexico, Panama City
  - Cevaxin La Chorrera, Panama City
  - INDICASAT Instituto de Investigaciones Científicas y Servicios de Alta Tecnología de Panamá, Panama City
- Asociacion Civil Selva Amazonica (ACSA), Iquitos, Peru
- Philippines (3):
  - De La Salle Health Sciences Institute- DLSUMC, Dasmariñas
  - Las Pinas Doctors Hospital, Las Piñas
  - Tropical Disease Foundation, Makati
- Ponce School of Medicine, Caimed Ctr, Ponce, Puerto Rico
- Thailand (4):
  - The Hospital for Tropical Diseases, Bangkok
  - Songklanagarind hospital, Hat Yai
  - Srinagarind Hospital, Muang
  - Research Institute for Health Science, Chiang Mai University, Muang

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 1595 enrolled participants (those who signed informed consent form [ICF]): 616 were index cases, 979 were household contacts (HHCs) identified from index cases. Of 616, 411 met the eligibility criteria for index case population (those who signed ICF and had a laboratory-confirmed dengue infection) and are reported below. Out of 979 HHCs, 128 were screen failures. Per plan, index cases were not included in any analysis and 851 randomized HHCs were included in the analysis.
Pre-assignment Details: HHCs included family members, acquaintances, co-workers, and community contacts, who were asymptomatic at screening (no clinical dengue symptoms). For safety assessments, although dosing stopped at Day 28, safety data through Day 50 were included in double-blind (DB) prophylactic phase due to drug's extended half-life (~10 days).
Groups:
- JNJ-64281802: High Dose Regimen: During the double-blind (DB) prophylactic dosing phase, HHC participants received loading dose of JNJ-64281802 400 milligrams (mg) tablet orally twice daily for 48 hours (Day 1 and 2) followed by maintenance dose of JNJ-64281802 150 mg tablet orally once daily for 26 days (from Day 3 to 28) in fed conditions. After Day 28, the prophylactic dosing phase was extended to Day 50 considering the long half-life (~10 days) of the study intervention. Participants then entered the follow-up phase and were followed up for safety up to Day 90 (end of trial).
- JNJ-64281802: Low Dose Regimen: During the DB prophylactic dosing phase, HHC participants received loading dose of JNJ-64281802 150 mg tablet orally twice daily for 48 hours (Day 1 and 2) followed by maintenance dose of JNJ-64281802 50 mg tablet orally once daily for 26 days (from Day 3 to 28) in fed conditions. After Day 28, the prophylactic dosing phase was extended to Day 50 considering the long half-life (~10 days) of the study intervention. Participants then entered the follow-up phase and were followed up for safety up to Day 90 (end of trial).
- Placebo: During the DB prophylactic dosing phase, HHC participants received placebo (matching to JNJ-64281802) tablet orally twice daily for 48 hours (Day 1 and 2) followed by orally once daily for 26 days (from Day 3 to 28) in fed conditions. After Day 28, the prophylactic dosing phase was extended to Day 50 considering the long half-life (~10 days) of the study intervention. Participants then entered the follow-up phase and were followed up for safety up to Day 90 (end of trial).
- Index Case Participants: Index case included all enrolled (on Day 1) participants who were with laboratory-confirmed dengue infection and contributed HHC participants. These index case participants were not randomized to receive study intervention.
Period: Overall Study
Arm/Group | JNJ-64281802: High Dose Regimen | JNJ-64281802: Low Dose Regimen | Placebo | Index Case Participants
Started | 283 | 283 | 285 | 411
Treated | 282 | 281 | 284 | 0
Participants Who Entered Into Follow-up Phase | 69 | 68 | 69 | 0
Completed | 247 | 250 | 252 | 411
Not Completed | 36 | 33 | 33 | 0
Not completed — Withdrawal by Subject | 13 | 12 | 14 | 0
Not completed — Adverse Event | 5 | 5 | 4 | 0
Not completed — Protocol-Specified Withdrawal Criterion Met | 5 | 1 | 4 | 0
Not completed — Non-Compliance With Study Drug | 2 | 3 | 3 | 0
Not completed — Physician Decision | 1 | 3 | 2 | 0
Not completed — Lost to Follow-up | 2 | 2 | 0 | 0
Not completed — Non-Compliance With Study Schedule | 1 | 1 | 1 | 0
Not completed — Protocol Violation | 2 | 0 | 1 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Site Terminated By Sponsor | 0 | 1 | 0 | 0
Not completed — Other | 3 | 3 | 3 | 0
Not completed — Randomized But Not Treated | 1 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: For randomized HHC participants: Safety analysis set included all randomized participants who received at least 1 dose of study intervention. For index case participants: Index case analysis set included all participants enrolled as an index case, with a laboratory-confirmed dengue virus (DENV) infection.
Groups:
- Total: Total of all reporting groups
Arm/Group | JNJ-64281802: High Dose Regimen | JNJ-64281802: Low Dose Regimen | Placebo | Index Case Participants | Total
Number analyzed (Participants) | 282 | 281 | 284 | 411 | 1258
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.8 (12.07) | 33.3 (11.67) | 34.7 (11.57) | 28.2 (16.54) | 32.3 (13.81)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 152 | 153 | 166 | 193 | 664
  Male | 130 | 128 | 118 | 217 | 593
  Undifferentiated | 0 | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 235 | 233 | 236 | 312 | 1016
  Not Hispanic or Latino | 47 | 47 | 47 | 91 | 232
  Unknown or Not Reported | 0 | 1 | 1 | 8 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 159 | 158 | 159 | 167 | 643
  Asian | 47 | 47 | 48 | 75 | 217
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 19 | 17 | 21 | 20 | 77
  White | 11 | 9 | 7 | 36 | 63
  More than one race | 15 | 16 | 18 | 20 | 69
  Unknown or Not Reported | 31 | 34 | 31 | 93 | 189
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 34 | 34 | 35 | 109 | 212
  Colombia | 132 | 129 | 131 | 110 | 502
  Mexico | 33 | 33 | 33 | 78 | 177
  Panama | 18 | 18 | 18 | 28 | 82
  Philippines | 23 | 23 | 23 | 28 | 97
  Thailand | 24 | 24 | 25 | 47 | 120
  Peru | 18 | 20 | 19 | 11 | 68

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Laboratory-confirmed Dengue Virus (DENV) Infection Between Baseline and the Last Day of Dosing + 1 Day Among Household Contacts (HHC) Participants With No Evidence of DENV Infection at Baseline
Description: Number of participants with DENV infection between baseline and the last day of dosing + 1 day among HHC participants with no evidence of DENV infection at baseline were reported. Presence of a laboratory-confirmed DENV infection was defined as a positive DENV ribonucleic acid (RNA) (assessed using a validated quantitative DENV reverse transcription polymerase chain reaction [RT-PCR]) or DENV non-structural protein 1 (NS1); assessed by enzyme-linked immunosorbent assay (ELISA) test result. A sample was considered positive for DENV RNA when the result was 'target detected' (when the result was above the limit of detection of the polymerase chain reaction [PCR] assay) or a sample was considered DENV NS1 positive if the qualitative DENV NS1 result was positive (quantitative DENV NS1 result greater than or equal to [>=] 11 relative units per milliliter [RU/mL]).
Time Frame: Baseline (DB prophylactic Day 1) up to last day of dosing + 1 day (up to DB prophylactic Day 29)
Population: Primary analysis set(PAS): all randomized participants who received at least 1 dose of study intervention, who had no evidence of DENV infection at baseline (based on target not detected [TND] results for DENV RNA assay and if available, negative/borderline result for NS1 protein assays) and with at least 1 result for DENV RNA or NS1 protein assay available post baseline up to and including last day of dosing + 1 day. As pre-planned, data collection and analysis was not performed for index case.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64281802: High Dose Regimen | JNJ-64281802: Low Dose Regimen | Placebo
Number analyzed (Participants) | 265 | 266 | 265
Participants | 2 | 2 | 6
Statistical Analysis 1: Comparison: JNJ-64281802: High Dose Regimen vs Placebo; The study was prematurely terminated before reaching the number of laboratory-confirmed DENV infections that were planned for the interim analysis. The 1-sided 20% significance level was described in the protocol as the significance level for proof-of-concept (PoC) when the planned interim analysis would have been performed; Test type: Superiority; p = 0.1409, Exact logistic regression model — One-sided p-value; P-value was obtained from an exact logistic regression model adjusted for stratification factor region (America, Asia); Odds Ratio (OR) = 67.3, 80% CI 1-sided [lower limit 15.2] — 1-sided odds-ratio and 80% CI were obtained from exact logistic regression model adjusted for region (America, Asia)
Statistical Analysis 2: Comparison: JNJ-64281802: Low Dose Regimen vs Placebo; The study was prematurely terminated before reaching the number of laboratory-confirmed DENV infections that were planned for the interim analysis. The 1-sided 20% significance level was described in the protocol as the significance level for PoC when the planned interim analysis would have been performed; Test type: Superiority; p = 0.1418, Exact logistic regression model — One-sided p-value; P-value was obtained from an exact logistic regression model adjusted for stratification factor region (America, Asia); Odds Ratio (OR) = 67.2, 80% CI 1-sided [lower limit 14.9] — 1-sided odds-ratio and 80% CI were obtained from exact logistic regression model adjusted for region (America, Asia)

2. Secondary Outcome: Number of Participants With Laboratory-confirmed Symptomatic DENV Infection Between Baseline and the Last Day of Dosing + 1 Day Among All HHC Participants (With or Without Evidence of DENV Infection at Baseline)
Description: Number of participants with laboratory-confirmed symptomatic DENV infection between baseline and last day of dosing + 1 day among all HHC participants (with/without evidence of DENV infection at baseline) were reported. Laboratory confirmed symptomatic DENV infection was defined as having at least 2 solicited systemic adverse events (AEs; retro-orbital pain, fever, arthralgia, headache, myalgia, rash, abdominal pain, nausea, fatigue, loss of appetite, vomiting, and diarrhea) of which at least 1 was a most common dengue symptom (retro-orbital pain, fever, arthralgia, headache, myalgia, rash), lasted for >=1 day and occurred within +/-2 days time window around positive PCR or NS1 test, between baseline and last day of dosing. Sample was considered positive for DENV RNA when result was 'target detected' (when result was above the limit of detection of PCR assay) or sample considered DENV NS1 positive if qualitative DENV NS1 result was positive (quantitative DENV NS1 result >=11 RU/mL).
Time Frame: Baseline (DB prophylactic Day 1) up to last day of dosing + 1 day (up to DB prophylactic Day 29)
Population: Complete analysis set: All participants included in PAS or secondary analysis set (SAS) (all randomized participants who received at least 1 dose of study intervention, had evidence of DENV infection [based on positive results for DENV RNA or NS1 protein assays at baseline] but without DENV signs and symptoms at baseline). As pre-planned, data collection and analysis was not performed for index case.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64281802: High Dose Regimen | JNJ-64281802: Low Dose Regimen | Placebo
Number analyzed (Participants) | 269 | 269 | 270
Participants | 1 | 3 | 8
Statistical Analysis 1: Comparison: JNJ-64281802: High Dose Regimen vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0192, Exact logistic regression model — One-sided p-value; P-value was obtained from an exact logistic regression model adjusted for stratification factor region (America, Asia); Odds Ratio (OR) = 87.8, 80% CI 1-sided [lower limit 58.1] — 1-sided odds-ratio and 80% CI were obtained from exact logistic regression model adjusted for region (America, Asia)
Statistical Analysis 2: Comparison: JNJ-64281802: Low Dose Regimen vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.1131, Exact logistic regression model — One-sided p-value; P-value was obtained from an exact logistic regression model adjusted for stratification factor region (America, Asia); Odds Ratio (OR) = 62.9, 80% CI 1-sided [lower limit 20] — 1-sided odds-ratio and 80% CI were obtained from exact logistic regression model adjusted for region (America, Asia)

3. Secondary Outcome: Number of Participants With Laboratory-confirmed Symptomatic DENV Infection Between Baseline and the Last Day of Dosing + 1 Day Among HHC Participants With No Evidence of DENV Infection at Baseline
Description: Number of participants with laboratory-confirmed symptomatic DENV infection between baseline and last day of dosing + 1 day among HHC participants with no evidence of DENV infection at baseline were reported. Laboratory confirmed symptomatic DENV infection was defined as having at least 2 solicited systemic AEs (retro-orbital pain, fever, arthralgia, headache, myalgia, rash, abdominal pain, nausea, fatigue, loss of appetite, vomiting, and diarrhea) of which at least 1 was a most common dengue symptom (retro-orbital pain, fever, arthralgia, headache, myalgia, and rash), lasted for >=1 day and occurred within a +/-2 days time window around the positive PCR or NS1 test, between baseline and the last day of dosing. A sample was considered positive for DENV RNA when the result was 'target detected' (when result was above the limit of detection of PCR assay) or sample was considered DENV NS1 positive if the qualitative DENV NS1 result was positive (quantitative DENV NS1 result >=11 RU/mL).
Time Frame: Baseline (DB prophylactic Day 1) up to last day of dosing + 1 day (up to DB prophylactic Day 29)
Population: PAS included all randomized participants who received at least 1 dose of study intervention, who had no evidence of DENV infection at baseline (based on TND] results for DENV RNA assay and, if available, a negative/borderline result for NS1 protein assays) and with at least 1 result for DENV RNA or NS1 protein assay available post baseline up to and including the last day of dosing + 1 day. As pre-planned, data collection and analysis was not performed for index case.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64281802: High Dose Regimen | JNJ-64281802: Low Dose Regimen | Placebo
Number analyzed (Participants) | 265 | 266 | 265
Participants | 0 | 2 | 5
Statistical Analysis 1: Comparison: JNJ-64281802: High Dose Regimen vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0302, Exact logistic regression model — One-sided p-value; P-value was obtained from an exact logistic regression model adjusted for stratification factor region (America, Asia); Odds Ratio (OR) = 85.4, 80% CI 1-sided [lower limit 62.6] — 1-sided odds-ratio and 80% CI were obtained from exact logistic regression model adjusted for region (America, Asia)
Statistical Analysis 2: Comparison: JNJ-64281802: Low Dose Regimen vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.2239, Exact logistic regression model — One-sided p-value; P-value was obtained from an exact logistic regression model adjusted for stratification factor region (America, Asia); Odds Ratio (OR) = 60.5, 80% CI 1-sided [lower limit -6.3] — 1-sided odds-ratio and 80% CI were obtained from exact logistic regression model adjusted for region (America, Asia)

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Serious AE was the AE resulting in any of following outcomes/deemed significant for any other reason: death; initial/prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs were defined as any AE occurring at or after initial administration of study intervention until the last study-related activity, or until the participant had been deemed lost to follow-up after demonstration of due diligence of follow up efforts. TEAEs included both serious and non-serious adverse events.
Time Frame: DB prophylactic phase: From start of study treatment (Day 1) up to visit Day 50, considering the long half-life (~10 days) of the study intervention; Follow-up phase: From visit Day 50 up to Day 90
Population: Safety analysis set included all randomized participants who received at least 1 dose of study intervention. As pre-planned, data collection and analysis was not performed for index case.
Measure: Count of Participants; unit: Participants
Groups:
- DB Prophylactic Phase: JNJ-64281802: High Dose Regimen: During the DB prophylactic dosing phase, HHC participants received loading dose of JNJ-64281802 400 mg tablet orally twice daily for 48 hours (Day 1 and 2) followed by maintenance dose of JNJ-64281802 150 mg tablet orally once daily for 26 days (from Day 3 to 28) in fed conditions. After Day 28, the prophylactic dosing phase was extended up to Day 50 considering the long half-life (~10 days) of the study intervention.
- DB Prophylactic Phase: JNJ-64281802: Low Dose Regimen: During the DB prophylactic dosing phase, HHC participants received loading dose of JNJ-64281802 150 mg tablet orally twice daily for 48 hours (Day 1 and 2) followed by maintenance dose of JNJ-64281802 50 mg tablet orally once daily for 26 days (from Day 3 to 28) in fed conditions. After Day 28, the prophylactic dosing phase was extended up to Day 50 considering the long half-life (~10 days) of the study intervention.
- DB Prophylactic Phase: Placebo: During the DB prophylactic dosing phase, HHC participants received placebo (matching to JNJ-64281802) tablet orally twice daily for 48 hours (Day 1 and 2) followed by orally once daily for 26 days (from Day 3 to 28) in fed conditions. After Day 28, the prophylactic dosing phase was extended up to Day 50 considering the long half-life (~10 days) of the study intervention.
- Follow-up Phase: JNJ-64281802: High Dose Regimen: After completion of DB prophylactic dosing phase, participants who received high dose of JNJ-64281802 in DB prophylactic dosing phase entered follow-up phase and were followed up for safety up to Day 90 (end of trial).
- Follow-up Phase: JNJ-64281802: Low Dose Regimen: After completion of DB prophylactic dosing phase, participants who received low dose of JNJ-64281802 in DB prophylactic dosing phase entered follow-up phase and were followed up for safety up to Day 90 (end of trial).
- Follow-up Phase: Placebo: After completion of DB prophylactic dosing phase, participants who received placebo (matching to JNJ-64281802) in DB prophylactic dosing phase entered follow-up phase and were followed up for safety up to Day 90 (end of trial).
Arm/Group | DB Prophylactic Phase: JNJ-64281802: High Dose Regimen | DB Prophylactic Phase: JNJ-64281802: Low Dose Regimen | DB Prophylactic Phase: Placebo | Follow-up Phase: JNJ-64281802: High Dose Regimen | Follow-up Phase: JNJ-64281802: Low Dose Regimen | Follow-up Phase: Placebo
Number analyzed (Participants) | 282 | 281 | 284 | 69 | 68 | 69
Participants
  TEAE | 169 | 162 | 176 | 13 | 8 | 8
  TESAE | 3 | 0 | 1 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Treatment-emergent (TE) Worst Grade (Grade 3 or 4) Abnormalities in Vital Signs
Description: Vital signs: pulse and blood pressure (systolic blood pressure[SBP]/diastolic blood pressure[DBP]). Abnormality grades determined per Division of Acquired Immunodeficiency Syndrome (DAIDS) for grading severity of adult and pediatric AEs: SBP(millimeters of mercury[mmHg]):Hypertension:Grade (G)1(mild):141-150, G2(moderate):greater than (>)150-155, G3(severe):>155; SBP(mmHg):Hypotension:G1(mild):85-89, G2(moderate):80 to less than (<)85, G3(severe):<80; DPB(mmHg):Hypertension:G1(mild):91-95, G2(moderate):>95-100, G3(severe):>100; Pulse(beats per minutes[bpm]):Tachycardia: G1(mild):>100-115, G2(moderate):>115-130, G3(severe):>130; Pulse(bpm):Bradycardia:G1(mild):50-54, G2(moderate):<50-45, G3(severe):<45. Any abnormality occurring at/after initial administration of study intervention until last study-related activity, or participant had been deemed lost to follow-up after demonstration of due diligence of follow up efforts was considered TE. Worst TE toxicity grade=highest grade reached.
Time Frame: From start of drug administration (DB prophylactic Day 1) up to Day 50
Population: Safety analysis set included all randomized participants who received at least 1 dose of study intervention. Here, 'N' (overall number of participants analyzed) refers to the number of participants evaluable for this outcome measure. Only parameter (SBP: Hypertension) in which at least 1 participant had data was reported. As pre-planned, data collection and analysis was not performed for index case.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64281802: High Dose Regimen | JNJ-64281802: Low Dose Regimen | Placebo
Number analyzed (Participants) | 255 | 258 | 259
Participants | 1 | 0 | 0

6. Secondary Outcome: Number of Participants With Treatment-emergent Abnormalities in Electrocardiogram (ECG) Parameters
Description: ECG variables: heart rate (HR), PR interval, RR interval, QRS interval, QT interval, and corrected QT (QTc) interval using both following correction methods: QT corrected according to Bazett's formula (QTcB), QT corrected according to Fridericia's formula (QTcF). Abnormalities were categorized as low or high. HR (bpm): low: < 45, high: >=120; PR Interval (milliseconds [ms]): low: <110, high: >=220; QRS interval (ms): high: >=120; QTcB and QTcF (ms): Borderline prolonged QT: 450< QTc <=480, 480 <QTc <=500, QTc >500. Any abnormality occurring at or after initial administration of study intervention until last study-related activity, or participant had been deemed lost to follow-up after demonstration of due diligence of follow up efforts was considered treatment emergent.
Time Frame: Day 28
Population: Safety analysis set included all randomized participants who received at least 1 dose of study intervention. Here, 'N' (overall number of participants analyzed) refers to the number of participants evaluable for this outcome measure; 'n' (number analyzed) signifies number of participants analyzed at specified rows. Only those parameters in which at least 1 participant had data was reported in this outcome measure. As pre-planned, data collection and analysis was not performed for index case.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64281802: High Dose Regimen | JNJ-64281802: Low Dose Regimen | Placebo
Number analyzed (Participants) | 252 | 254 | 258
Participants
  Heart Rate: Abnormally Low (<45) | 1 | 0 | 0
  PR Interval, Aggregate: Abnormally High (>=220): number analyzed (Participants) | 252 | 254 | 257
  PR Interval, Aggregate: Abnormally High (>=220) | 0 | 1 | 2
  PR Interval, Aggregate: Abnormally Low (<110): number analyzed (Participants) | 252 | 254 | 257
  PR Interval, Aggregate: Abnormally Low (<110) | 1 | 0 | 2
  QTcB Interval, Aggregate: Borderline prolonged QT (450< QTc <=480) | 1 | 2 | 0
  QTcF Interval, Aggregate: Borderline prolonged QT (450< QTc <=480) | 0 | 1 | 0
  QRS Duration, Aggregate: Abnormally High (>=120) | 1 | 1 | 0

7. Secondary Outcome: Number of Participants With Treatment-emergent Worst Grade (Grade 3 or 4) Abnormalities in Laboratory Parameters
Description: Number of participants with treatment-emergent worst grade (Grade 3 or 4) abnormalities in laboratory parameters were reported. Laboratory assessments included clinical chemistry, hematology and urinalysis. Abnormality criterions were based on DAIDS: Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening. Any abnormality occurring at or after initial administration of study intervention until the last study-related activity, or until the participant had been deemed lost to follow-up after demonstration of due diligence of follow up efforts was considered treatment emergent.
Time Frame: From start of drug administration (DB prophylactic Day 1) up to Day 50
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64281802: High Dose Regimen | JNJ-64281802: Low Dose Regimen | Placebo
Number analyzed (Participants) | 271 | 270 | 278
Participants
  Hematology: Hemoglobin, Low: Grade 3: number analyzed (Participants) | 266 | 270 | 273
  Hematology: Hemoglobin, Low: Grade 3 | 1 | 1 | 3
  Hematology: Hemoglobin, Low: Grade 4: number analyzed (Participants) | 266 | 270 | 273
  Hematology: Hemoglobin, Low: Grade 4 | 1 | 2 | 0
  Hematology: Activated partial thromboplastin time (APTT), High: Grade 3 | 1 | 0 | 0
  Hematology: APTT, High: Grade 4 | 1 | 0 | 2
  Hematology: Prothrombin time (PT), High: Grade 3 | 1 | 0 | 0
  Hematology: PT, High: Grade 4 | 1 | 1 | 4
  Hematology: Platelets, Decrease: Grade 3: number analyzed (Participants) | 266 | 270 | 273
  Hematology: Platelets, Decrease: Grade 3 | 0 | 0 | 3
  Chemistry: Hyperglycemia: Grade 3 | 10 | 17 | 14
  Chemistry: Hypoglycemia: Grade 3 | 1 | 3 | 1
  Chemistry: Hypoglycemia: Grade 4 | 1 | 0 | 0
  Chemistry: Triglycerides (Fasting), High: Grade 3 | 2 | 2 | 1
  Chemistry: Cholesterol, High: Grade 3 | 22 | 17 | 20
  Chemistry: Low density lipoprotein (Fasting), High: Grade 3: number analyzed (Participants) | 264 | 261 | 271
  Chemistry: Low density lipoprotein (Fasting), High: Grade 3 | 4 | 3 | 8
  Chemistry: Hypernatremia: Grade 4 | 1 | 0 | 0
  Chemistry: Creatine Kinase, High: Grade 3 | 2 | 4 | 4
  Chemistry: Creatine Kinase, High: Grade 4 | 3 | 2 | 0
  Chemistry: Alanine aminotransferase or Serum glutamic pyruvic transaminase (SGPT), High: Grade 3 | 0 | 1 | 0
  Chemistry: Uric Acid, High: Grade 3 | 0 | 1 | 0
  Chemistry: Hyperkalemia: Grade 3 | 0 | 1 | 0
  Chemistry: Hypokalemia: Grade 3 | 1 | 0 | 2
  Chemistry: Gamma Glutamyl Transferase, High: Grade 3 | 1 | 0 | 0
  Chemistry: Amylase (Pancreatic), High: Grade 4: number analyzed (Participants) | 242 | 241 | 249
  Chemistry: Amylase (Pancreatic), High: Grade 4 | 1 | 0 | 0
  Chemistry: Hypophosphatemia: Grade 3 | 2 | 0 | 0
  Chemistry: Aspartate aminotransferase or Serum glutamic-oxaloacetic transaminase, High: Grade 3 | 0 | 1 | 0
  Chemistry: Hyperbilirubinemia: Grade 4 | 1 | 0 | 0
  Chemistry: Hypercalcemia: Grade 3 | 0 | 1 | 0
  Chemistry: Hypocalcemia: Grade 4 | 0 | 1 | 0
  Chemistry: Lipase, High: Grade 3 | 2 | 0 | 0
  Urinalysis: Protein, High: Grade 3: number analyzed (Participants) | 254 | 262 | 260
  Urinalysis: Protein, High: Grade 3 | 0 | 1 | 2
  Urinalysis: Glycosuria: Grade 3: number analyzed (Participants) | 254 | 262 | 260
  Urinalysis: Glycosuria: Grade 3 | 2 | 0 | 2

8. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Physical Examinations
Description: Number of participants with abnormalities in physical examination parameters (head/neck/thyroid, eyes/ears/nose/throat, respiratory, cardiovascular, lymph nodes, abdomen, skin, musculoskeletal, and neurological) were reported based on investigator's discretion.
Time Frame: Day 50
Population: Safety analysis set included all randomized participants who received at least 1 dose of study intervention. Here, 'N' (overall number of participants analyzed) refers to the number of participants evaluable for this outcome measure. As pre-planned, data collection and analysis was not performed for index case.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64281802: High Dose Regimen | JNJ-64281802: Low Dose Regimen | Placebo
Number analyzed (Participants) | 248 | 250 | 255
Participants | 7 | 9 | 13

9. Secondary Outcome: Plasma Concentrations of JNJ-64281802
Description: Plasma concentrations of JNJ-64281802 were reported. Plasma samples were analyzed using liquid chromatography-tandem mass spectrometry (LC-MS/MS) method.
Time Frame: Pre-dose on Day 1; post-dose on Days 3, 5,9, 13, 21, and 28 ; Days 40, 50, and 90
Population: Pharmacokinetic analysis set included all participants who received at least 1 dose of study intervention and who had at least 1 plasma concentration data value after dosing. Here 'N' (overall number of participants analyzed) refers to the number of participants evaluable for this outcome measure, 'n' (number analyzed) refers to all participants evaluable at specified time points. Data for this outcome measure was planned to be collected and analyzed for specified arms only.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | JNJ-64281802: High Dose Regimen | JNJ-64281802: Low Dose Regimen
Number analyzed (Participants) | 267 | 268
Nanograms per milliliter (ng/mL)
  Pre-dose on Day 1 | 1.9 (31.52) | 4.2 (69.03)
  Post-dose on Day 3: number analyzed (Participants) | 51 | 49
  Post-dose on Day 3 | 4233.5 (1534.79) | 1777.1 (732.09)
  Post-dose on Day 5: number analyzed (Participants) | 261 | 255
  Post-dose on Day 5 | 2735.0 (1370.95) | 1037.1 (505.93)
  Post-dose on Day 9: number analyzed (Participants) | 258 | 264
  Post-dose on Day 9 | 2583.1 (1311.77) | 909.1 (469.41)
  Post-dose on Day 13: number analyzed (Participants) | 249 | 258
  Post-dose on Day 13 | 2657.4 (1380.73) | 865.8 (439.79)
  Post-dose on Day 21: number analyzed (Participants) | 248 | 254
  Post-dose on Day 21 | 2649.4 (1606.28) | 846.9 (495.83)
  Post-dose on Day 28: number analyzed (Participants) | 248 | 249
  Post-dose on Day 28 | 2614.1 (1653.06) | 816.1 (535.34)
  Day 40: number analyzed (Participants) | 245 | 248
  Day 40 | 1194.8 (858.11) | 325.4 (238.77)
  Day 50: number analyzed (Participants) | 246 | 245
  Day 50 | 640.2 (543.84) | 165.4 (143.87)
  Day 90: number analyzed (Participants) | 65 | 61
  Day 90 | 57.3 (82.76) | 12.0 (18.82)

ADVERSE EVENTS:
Time Frame: All Cause Mortality: DB prophylactic phase: From randomization (pre-dose, DB prophylactic Day 1) up to Day 50, Follow up phase: From Day 50 up to end of trial (Day 90); Serious and Other AEs: DB prophylactic phase: From start of study treatment (DB prophylactic Day 1) up to Day 50, Follow-up phase: From Day 50 up to End of trial (Day 90)
Description: All Cause Mortality: Randomized analysis set included all HHC participants who were randomized in the study. Serious and Other AEs: Safety analysis set included all randomized participants who received at least 1 dose of study intervention. Per plan, safety data collection and analysis was not performed for index case. Although dosing stopped at Day 28, safety data through Day 50 were included in the DB prophylactic phase due to the drug's extended half-life (~10 days).
Groups:
- DB Prophylactic Phase: Placebo: During the DB prophylactic dosing phase, HHC participants received placebo (matching JNJ-64281802) tablet orally twice daily for 48 hours (Day 1 and 2) followed by once daily for 26 days (from Day 3 to 28) in fed conditions. After Day 28, the prophylactic dosing phase was extended up to Day 50 considering the long half-life (~10 days) of the study intervention.
Arm/Group | DB Prophylactic Phase: JNJ-64281802: High Dose Regimen | DB Prophylactic Phase: JNJ-64281802: Low Dose Regimen | DB Prophylactic Phase: Placebo | Follow-up Phase: JNJ-64281802: High Dose Regimen | Follow-up Phase: JNJ-64281802: Low Dose Regimen | Follow-up Phase: Placebo
All-Cause Mortality (participants affected / at risk) | 1/283 | 0/283 | 0/285 | 0/69 | 0/68 | 0/69
Serious Adverse Events (participants affected / at risk) | 3/282 | 0/281 | 1/284 | 0/69 | 0/68 | 0/69
Other Adverse Events (participants affected / at risk) | 107/282 | 106/281 | 109/284 | 9/69 | 6/68 | 8/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Prophylactic Phase: JNJ-64281802: High Dose Regimen (N=282) | DB Prophylactic Phase: JNJ-64281802: Low Dose Regimen (N=281) | DB Prophylactic Phase: Placebo (N=284) | Follow-up Phase: JNJ-64281802: High Dose Regimen (N=69) | Follow-up Phase: JNJ-64281802: Low Dose Regimen (N=68) | Follow-up Phase: Placebo (N=69)
Angina Unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertensive Heart Disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Crush Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Hypertensive Crisis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Prophylactic Phase: JNJ-64281802: High Dose Regimen (N=282) | DB Prophylactic Phase: JNJ-64281802: Low Dose Regimen (N=281) | DB Prophylactic Phase: Placebo (N=284) | Follow-up Phase: JNJ-64281802: High Dose Regimen (N=69) | Follow-up Phase: JNJ-64281802: Low Dose Regimen (N=68) | Follow-up Phase: Placebo (N=69)
Abdominal Pain (Gastrointestinal disorders) | 16 | 13 | 20 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 35 | 23 | 23 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 18 | 21 | 24 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 8 | 8 | 15 | 1 | 0 | 0
Fatigue (General disorders) | 16 | 25 | 26 | 1 | 1 | 0
Pyrexia (General disorders) | 22 | 25 | 39 | 4 | 3 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 7 | 6 | 2 | 4 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 6 | 9 | 20 | 0 | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 19 | 15 | 20 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 17 | 23 | 3 | 3 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 15 | 25 | 1 | 1 | 0
Headache (Nervous system disorders) | 54 | 61 | 67 | 4 | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 4 | 3 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/94/NCT05201794/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-21): https://cdn.clinicaltrials.gov/large-docs/94/NCT05201794/SAP_001.pdf